CLINICAL TRIAL: NCT00279825
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Compare IPX054 200 mg and 250 mg to CD-LD IR 200 (2x100) mg Tablets and CD-LD CR 200 mg Tablet in Subjects With Parkinson's Disease
Brief Title: Comparison of IPX054, IR Carbidopa-Levodopa, and CR Carbidopa-Levodopa in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IPX054-B05-01
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2017-01

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Other): Subjects take 1 tablet of IPX054 200 mg, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR Placebo. In Second treatment, subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR Placebo. In Third treatment, subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR and 1 tablet of CD-LD CR Placebo. In Fourth treatment, subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR.
  Interventions: Drug: IPX054 200 mg; Drug: IPX054 250 mg; Drug: CD-LD IR; Drug: CD-LD CR; Drug: IPX054 200 mg Placebo; Drug: IPX054 250 mg Placebo; Drug: CD-LD IR Placebo; Drug: CD-LD CR Placebo
- Sequence 2 (Other): Subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR Placebo. In Second treatment, subjects take 1 tablet of IPX054 200 mg, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR Placebo. In Third treatment, subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR. In Fourth treatment, subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR and 1 tablet of CD-LD CR Placebo.
  Interventions: Drug: IPX054 200 mg; Drug: IPX054 250 mg; Drug: CD-LD IR; Drug: CD-LD CR; Drug: IPX054 200 mg Placebo; Drug: IPX054 250 mg Placebo; Drug: CD-LD IR Placebo; Drug: CD-LD CR Placebo
- Sequence 3 (Other): Subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR and 1 tablet of CD-LD CR Placebo. In Second treatment, subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR. In Third treatment, subjects take 1 tablet of IPX054 200 mg, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR Placebo. In Fourth treatment, subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR Placebo.
  Interventions: Drug: IPX054 200 mg; Drug: IPX054 250 mg; Drug: CD-LD IR; Drug: CD-LD CR; Drug: IPX054 200 mg Placebo; Drug: IPX054 250 mg Placebo; Drug: CD-LD IR Placebo; Drug: CD-LD CR Placebo
- Sequence 4 (Other): Subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR. In Second treatment, subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR and 1 tablet of CD-LD CR Placebo. In Third treatment, subjects take 1 tablet of IPX054 200 mg Placebo, 1 tablet of IPX054 250 mg, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR Placebo. In Fourth treatment, subjects take 1 tablet of IPX054 200 mg, 1 tablet of IPX054 250 mg Placebo, 2 tablets of CD-LD IR Placebo and 1 tablet of CD-LD CR Placebo.
  Interventions: Drug: IPX054 200 mg; Drug: IPX054 250 mg; Drug: CD-LD IR; Drug: CD-LD CR; Drug: IPX054 200 mg Placebo; Drug: IPX054 250 mg Placebo; Drug: CD-LD IR Placebo; Drug: CD-LD CR Placebo

INTERVENTIONS:
Drug: IPX054 200 mg — IPX054 tablet containing 50 mg carbidopa and 200 mg levodopa
Drug: IPX054 250 mg — IPX054 tablet containing 62.5 mg carbidopa and 250 mg levodopa
Drug: CD-LD IR — Active comparator containing 25 mg carbidopa and 100 mg levodopa
  Other Names: Carbidopa-levodopa immediate-release tablets
Drug: CD-LD CR — Active comparator containing 50 mg carbidopa and 200 mg levodopa
  Other Names: Carbidopa-levodopa controlled-release tablets
Drug: IPX054 200 mg Placebo — Placebo to match IPX054 200 mg
Drug: IPX054 250 mg Placebo — Placebo to match IPX054 250 mg
Drug: CD-LD IR Placebo — Placebo to match CD-LD IR
Drug: CD-LD CR Placebo — Placebo to match CD-LD CR

SUMMARY:
The objective of this study is to compare the pharmacokinetics and pharmacodynamics of IPX054, carbidopa-levodopa immediate-release tablets, and carbidopa-levodopa controlled-release tablets in subjects with idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
IPX054 contains two different drugs called levodopa and carbidopa in one tablet.

* levodopa turns into a material called 'dopamine' in your brain. The dopamine helps to improve the symptoms of your Parkinson's disease.
* carbidopa belongs to a group of medicines called 'aromatic amino acid decarboxylase inhibitors'. It helps levodopa work more effectively by slowing the speed at which levodopa is broken down in your body.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease.
* Currently being treated with immediate-release or controlled-release carbidopa-levodopa and not requiring more than 200 mg levodopa per dose.
* Must experience "wearing OFF" between doses of medication.

Exclusion Criteria:

* Diagnosed with atypical parkinsonism.
* Allergic or non-responsive to previous carbidopa-levodopa therapy.
* Active or history of narrow-angle or wide-angle glaucoma.
* History of seizure or epilepsy, or is currently taking an anti-convulsant for treatment of seizures.
* Treatment with any neuroleptic agent, including atypical neuroleptics, within the previous 12 months.
* Treatment with any dopaminergic blocking agent within the previous 3 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Alternate tapping of keys | single dose

SECONDARY OUTCOMES:
Timed walking | single dose
Tremor score | single dose
Dyskinesia rating scale | single dose

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (2):
- United States (2):
  - Quest Research Institute, Bingham Farms, Michigan
  - Oregon Health Sciences University - Parkinson's Center of Oregon, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No